CLINICAL TRIAL: NCT02385487
Title: Inflammation in Type 2 Myocardial Infarction
Status: Withdrawn | Type: Observational
Why Stopped: Logistics and feasibility
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: S14-01349
Record Dates: First submitted 2015-02-26; First posted 2015-03-11 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Myocardial Infarction; Inflammation; Critical Illness
Keywords: Myocardial Infarction; Inflammation; Critical Illness; Necrosis; Sepsis; Respiratory Insufficiency; Myocardial Ischemia; Cardiovascular Diseases; Heart Diseases; Vascular Diseases
MeSH Terms: conditions — Myocardial Infarction; Inflammation; Critical Illness; Necrosis; Sepsis; Respiratory Insufficiency; Myocardial Ischemia; Cardiovascular Diseases; Heart Diseases; Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Critical illness and type 2 MI: Critically ill adults with abnormal serum troponin I during hospitalization for critical illness.
- Critical illness without type 2 MI: Critically ill adults without an elevation in troponin I complicating critical illness.

SUMMARY:
Type 2 myocardial infarction (MI) is defined as myocardial necrosis that results from an imbalance of myocardial oxygen supply and demand. Although type 2 MI is highly prevalent in patients with critical illness and strongly associated with mortality, the pathophysiology remains poorly understood. Inflammation is central to the development of atherosclerosis, plaque rupture, and other subtypes of MI, but the role of inflammation in type 2 MI and myocardial necrosis has not been defined. The investigators aim to to delineate the mechanistic role of inflammation in myocardial necrosis and type 2 MI complicating critical medical illness.

ELIGIBILITY:
Inclusion Criteria:

* ≥21 years of age
* admitted to the Medical Intensive or Coronary Care Units
* sepsis or respiratory failure
* clinically indicated troponin measurement within 24 hours of ICU admission

Exclusion Criteria:

* unstable angina or Type 1 MI
* percutaneous or surgical coronary revascularization within 7 days
* heart failure exacerbation
* primary valvular disorder
* aortic dissection
* infiltrative heart disease or hypertrophic cardiomyopathy
* myocarditis
* pulmonary embolism
* electrocardiogram with >1mm ST segment elevation in two consecutive leads
* serum cardiac troponin >99th percentile URL but no clear rise or fall pattern
* history of chronic inflammatory disease
* use of therapeutic-dose anticoagulants / antiplatelet agents other than aspirin
* pregnant or incarcerated
* enrolled in a competing study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults admitted to the Medical Intensive or Coronary Care Units (MICU or CCU)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Leukocyte-platelet aggregates | Day 1

SECONDARY OUTCOMES:
Leukocyte-platelet aggregates | Day 10
  Participants will be followed for the duration of hospital stay, an expected average of 10 days.
Monocyte-platelet aggregates | Day 1
Monocyte-platelet aggregates | Day 10
  Participants will be followed for the duration of hospital stay, an expected average of 10 days.
Neutrophil-platelet aggregates | Day 1
Neutrophil-platelet aggregates | Day 10
  Participants will be followed for the duration of hospital stay, an expected average of 10 days.

OTHER OUTCOMES:
EndoPAT score | Day 1
EndoPAT score | Day 10
  Participants will be followed for the duration of hospital stay, an expected average of 10 days.
surface L-selectin | Day 1
surface L-selectin | Day 10
  Participants will be followed for the duration of hospital stay, an expected average of 10 days.
soluble L-selectin | Day 1
soluble L-selectin | Day 10
  Participants will be followed for the duration of hospital stay, an expected average of 10 days.
surface CD11b | Day 1
surface CD11b | Day 1
  Participants will be followed for the duration of hospital stay, an expected average of 10 days.

CONTACTS AND LOCATIONS:
Overall Officials: Binita Shah, MD, MS, Principal Investigator — NYU School of Medicine
Locations (1):
- Bellevue Hospital Center, New York, New York, United States